CLINICAL TRIAL: NCT00443378
Title: Computer Assisted Rx Education for HIV-Positives: CARE+
Acronym: CARE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Ann Kurth, CNM, PhD, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 04-3810-C 01
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: computer counseling; HIV; antiretroviral adherence; sexual behavior; prevention with positives; HIV seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Arm 1, "CARE+ arm" is the study arm that receives the CARE+ computer intervention.
  Interventions: Behavioral: CARE+
- 2 (No Intervention): Arm 2, the control arm, is the study arm that receives computerized risk assessment only.
  Interventions: Behavioral: CARE+

INTERVENTIONS:
Behavioral: CARE+ — CARE+ is a .NET based application on tablet computers that comprises risk assessment, medication monitoring, tailored feedback, stage-based skills-building videos, motivational interviewing counseling, an integrated health promotion plan, and printout with referrals. Evidence-based approaches (pharmacist education, self-efficacy/importance scaling exercises, and consequence-framing) are incorporated.

SUMMARY:
This study evaluates an interactive computer counseling tool to help HIV-positive individuals develop an integrated health promotion plan incorporating antiretroviral (ART) adherence and HIV transmission risk reduction. We hypothesize that evidence-based counseling for ART adherence support and for HIV transmission risk reduction can be delivered effectively in a self-administered computer tool.

DETAILED DESCRIPTION:
Strict adherence to ART regimens is necessary for viral suppression and to avoid development of viral resistance, yet average ART adherence among HIV-positive individuals in North America is only 55%. Focused prevention efforts are key to reduce secondary HIV transmission to sexual and needle-sharing partners, yet many HIV patients do not receive counseling about these behaviors from their providers. Despite the global pandemic and a rising HIV incidence among some US populations, few health promotion interventions have integrated ART adherence with transmission risk reduction for people living with HIV. Most of the efficacious adherence or prevention interventions to date are not practical to scale up, as they require intense staff training and quality assurance and can be delivered to relatively few individuals at any one time.

An interactive health communication tool promises the possibility of a cost-effective adjunct to existing human-delivered counseling, or a stand-alone intervention when no other counseling would otherwise be offered.

This RCT of one such tool -- CARE+ --will provide empiric evidence of the benefits and limits of a computerized health promotion intervention to integrate ART adherence with transmission prevention for individuals with HIV. CARE+ is a .NET based application on tablet computers that comprises risk assessment, medication monitoring, tailored feedback, stage-based skills-building videos, motivational interviewing counseling, an integrated health promotion plan, and printout with referrals. Evidence-based approaches (pharmacist education, self-efficacy/importance scaling exercises, and consequence-framing) are incorporated.

Comparison: The CARE+ longitudinal RCT compares clinical and behavioral outcomes of CARE+ users to a control arm which assesses audio computer-assisted self-interview risk behaviors only. Participants were recruited and enrolled at two study sites, 1) an urban outpatient HIV clinic and 2) a community based AIDS Service Organization.

Aim 1: Identify common elements of adherence and transmission behaviors, health communication needs, and technology attitudes (n=30 interviews); incorporate into CARE+ and test software usability (n=30). Aim 2: Randomized clinical trial of HIV-positive adults on ART. Arm 1: CARE+ (n=120); Arm 2: computer risk assessment only (n=120). Arms 1 and 2 perform baseline, 3-, 6-, and 9-month session. Compare outcomes: a) ART adherence by plasma HIV viral load, CD4, self-report and b) HIV transmission sexual risk behaviors at follow-up. Aim 3: Provide data for HIV transmission dynamics impact modeling.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* currently taking highly active antiretroviral medication

Exclusion Criteria:

* unable to understand spoken English
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
HIV-1 viral load | 0,3,6 and 9 months
Self-reported 30-day visual analogue scale and 7-day missed dose report (adherence) | 0,3,6 and 9 months
Self-reported unprotected sex w/ nonconcordant partner (HIV transmission risk) | 0,3,6 and 9 months
CD4 cell count | 0,3,6 and 9 months

SECONDARY OUTCOMES:
Compare self-report to pharmacy refill and other chart data at 0,3,6,9 months | 0,3,6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kurth, CNM, PhD, Principal Investigator — University Washington, School of Nursing
Locations (2):
- United States (2):
  - Lifelong AIDS Alliance, Seattle, Washington
  - Madison Clinic, Harborview Medical Center, Seattle, Washington